CLINICAL TRIAL: NCT04527315
Title: Assessment of ICU and Non-ICU Survivors: A Creation of a COVID Survivorship Database
Brief Title: COVID-19 Survivorship Registry
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 20-00909
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood will be tested for cytokine levels, inflammatory markers and genetics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 ICU Patients
  Interventions: Other: Questionnaires
- Control
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Various questionnaires will be used to assess short and long-term impacts of depression, anxiety, and other indicators of overall mental health and quality of life

SUMMARY:
COVID-19 is associated with acute pulmonary and cardiac injury. To better understand the degree and severity of cardiopulmonary injury as well as short and long-term sequelae of COVID-19 infection, this study will perform longitudinal study in patients who had recent known diagnosis of COVID-19.

DETAILED DESCRIPTION:
The objectives for this study include providing structural and function information about lung and heart using chest imaging, MRI, Echo, Spirometry, and blood markers in order to assess severity of cardiopulmonary injury and short- and long-term sequelae of COVID-19 infection as well as assess indicators of mental health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* have tested positive for SARS-CoV-2 and discharged from the ICU or,
* have tested positive for SARS-CoV-2 and have been discharged from hospital or,
* have tested positive for SARS-CoV-2 but was NOT hospitalized
* ages 18 and over, and
* competent and willing to sign informed consent and comply to all aspects of the protocol

CONTROL Inclusion Criteria

* No clinical history of COVID-19,
* No active clinical symptoms indicative of possible COVID-19,
* Ages 18 and over,
* competent and willing to sign informed consent and comply to all aspects of the protocol

Exclusion Criteria:

• Participants cannot sign consent

Any individual who meets any of the following criteria will be excluded from participation to the MRI or x-ray portion of the study:

* Participants who are pregnant or currently trying to get pregnant
* Participants unable to comply with any portion of the protocol (i.e. removing metals prior to entering the MRI scan room) or who have contraindications to MRI scanning (i.e., non-MRI-conditional pacemakers/defibrillators, pregnancy, ferromagnetic implants such as aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
* Persistent symptoms related to COVID-19 (in which case the patient may be re-screened later) As is done for all patients undergoing clinical MRI in our department, each patient will be screened for contraindications to MRI with a routine questionnaire prior to scanning.

CONTROL Exclusion Criteria

Patients with any of the following are excluded from as controls:

* Pace maker
* Poorly controlled diabetes
* Poorly controlled Restrictive lung disease
* Heart failure
* Parkinson's Disease
* Hypertension
* Any diagnosis or history of autonomic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have had a positive COVID-19 test, but were not hospitalized/admitted will also be identified and eligible to participate in the study. Age and sex matched controls will also be recruited from those with no clinical history of COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-07-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Level of Inflammatory Markers | Up to 12 months
  Inflammatory markers include D-dimer, ferritin, and CRP measurements

SECONDARY OUTCOMES:
Score on St. George's Shortness of Breath Questionnaire (SGSQ) | Up to 12 months
  Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Score on Short Form Zarit Burden Interview (ZBI-12) | Up to 12 months
  Short form ZBI-12 validated as screening tool in advanced illness including dementia and cancer. Total ZBI-12 score: summation of 12 items (0 to 4 points per item, total score range 0 to 48). The higher the score, the higher the burden.

CONTACTS AND LOCATIONS:
Overall Officials: Rany Condos, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to covid-19survivorship@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.